CLINICAL TRIAL: NCT01800058
Title: Prognostic Value of the Levels of Circulating Tumor Cells (CTCs) in Peripheral Blood in Patients With Prostate Cancer at High Risk (Clinical Stages IIB-III) Treated Radically With Radiotherapy and Hormone Therapy.
Brief Title: Circulating Tumor Cells in High-Risk Prostate Cancer Treated With High-dose Radiotherapy and Hormone Therapy
Status: Completed | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Other Study IDs: CaPr-RTCTC-01/PI 197
Record Dates: First submitted 2013-02-18; First posted 2013-02-27 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Patients With High-risk Prostate Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prospective analysis of biological material from samples of peripheral blood (PB) of patients with high risk prostate cancer treated with dose escalation RT combined with androgen deprivation (AD)
  The sampling of PB for detection of CTCs was performed at 4 timepoints:
  * Before starting any treatment
  * Prior to the start of RT and after neoadjuvant AD
  * At the end of RT (1-3 months)
  * 6-12 months following the end of RT in patients with 0 CTCs in the 1º determination and positive CTCs in the 2º or 3º determination.
  A cut off of 0 vs ≥ 1 CTC/7.5 mL blood was defined as a threshold for negative versus positive CTCs status.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Circulating prostatic tumor cells in the peripheral blood: Patients that satisfy inclusion criteria, and after signing informed consent, will extract 1 blood sample (7.5 mL):
  1. prior to any treatment;
  2. following AD and prior to RT; and
  3. following the end of RT (1-3 months afterwards).
  4. six to twelve months following the end of RT in those patients with 0 CTCs in the first determination and positive CTCs in the second or third determination
  The quantification of CTC in blood samples will be done with the CellSearch® system.

SUMMARY:
The detection and quantification of Circulating tumor cells CTCs in peripheral blood of patients with prostate adenocarcinoma may be useful at least for:

Getting a correct stratification of patients with high-risk prostate cancer (PCa).

Set the prognosis at baseline. Evaluate the response to different treatments (predictive value and monitoring).

Establish individualized therapies.

DETAILED DESCRIPTION:
Prospective analysis of biologic samples from peripheral blood of 65 patients with localized high-risk PCa (NCCN 2011) treated with RTC-3D-IMRT combined with AD.

Following the sign of the informed consent of the patient, the blood samples will be analyzed for CTCs using an immunomagnetic method based on the CellSearch system (Veridex), in 4 periods of time:

1. prior to any treatment;
2. following AD and prior to RT; and
3. following the end of RT (1-3 months afterwards).
4. six to twelve months following the end of RT in those patients with 0 CTCs in the first determination and positive CTCs in the second or third determination

Comparison between the expression of CTCs in peripheral blood before and following AD and RT will be performed. The quantification of the CTCs obtained in these phases of treatment will be correlated with the treatment results in terms of biochemical failure according to Phoenix definition, distant metastasis rate and overall survival to identify a significant prognostic relationship and to determine the potential effect of the treatment in the number of CTCs Our working group will include 65 patients because the amount is based on routine clinical activity can be safely enrolled in the project development time by the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 with capacity to give informed consent.
* Patients with histologically confirmed prostate cancer.
* Patients with a high risk factor: PSA> 20 ng / ml, Gleason 8-10 and / or stage T3a-b, N0M0 (NCCN 2011, stage IIB-III AJCC classification 2010). Staging by: Histology-Gleason score-, PSA, TR, ECO TR, CT, MRI.
* Patients who accept radical treatment with radiotherapy.
* Patients who give written informed consent to participate in the study

Exclusion Criteria:

* Any patient diagnosed with prostate cancer, which does not meet the prerequisites.
* Any patients with another malignancy diagnosed in the past 5 years (except basal cell or squamous cell carcinoma of skin).
* Any patient who has prostate biopsy performed 7 days prior to study entry.
* Patients who have received prior treatment with hormonal therapy, chemotherapy or radiotherapy.
* Patients with PSA> 100 ng / ml.
* Any situation or condition of the patient which in the opinion of the investigator, advised against participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with prostate cancer at high risk (NCCN 2011), AJCC stage IIB-III, treated with 3D-CRT, IMRT dose escalation (with androgen deprivation (DA))
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Almudena Zapatero, MD, PhD, PI, Principal Investigator — Radiation Oncology Department_Hospital Universitario de La Princesa
Locations (3):
- Spain (3):
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

REFERENCES:
- [Background] Damber JE, Aus G. Prostate cancer. Lancet. 2008 May 17;371(9625):1710-21. doi: 10.1016/S0140-6736(08)60729-1. PMID 18486743
- [Background] Zelefsky MJ, Yamada Y, Fuks Z, Zhang Z, Hunt M, Cahlon O, Park J, Shippy A. Long-term results of conformal radiotherapy for prostate cancer: impact of dose escalation on biochemical tumor control and distant metastases-free survival outcomes. Int J Radiat Oncol Biol Phys. 2008 Jul 15;71(4):1028-33. doi: 10.1016/j.ijrobp.2007.11.066. Epub 2008 Feb 14. PMID 18280056
- [Background] Kuban DA, Tucker SL, Dong L, Starkschall G, Huang EH, Cheung MR, Lee AK, Pollack A. Long-term results of the M. D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):67-74. doi: 10.1016/j.ijrobp.2007.06.054. Epub 2007 Aug 31. PMID 17765406
- [Background] Roach M 3rd, Bae K, Speight J, Wolkov HB, Rubin P, Lee RJ, Lawton C, Valicenti R, Grignon D, Pilepich MV. Short-term neoadjuvant androgen deprivation therapy and external-beam radiotherapy for locally advanced prostate cancer: long-term results of RTOG 8610. J Clin Oncol. 2008 Feb 1;26(4):585-91. doi: 10.1200/JCO.2007.13.9881. Epub 2008 Jan 2. PMID 18172188
- [Background] Horwitz EM, Bae K, Hanks GE, Porter A, Grignon DJ, Brereton HD, Venkatesan V, Lawton CA, Rosenthal SA, Sandler HM, Shipley WU. Ten-year follow-up of radiation therapy oncology group protocol 92-02: a phase III trial of the duration of elective androgen deprivation in locally advanced prostate cancer. J Clin Oncol. 2008 May 20;26(15):2497-504. doi: 10.1200/JCO.2007.14.9021. Epub 2008 Apr 14. PMID 18413638
- [Background] Shaffer DR, Leversha MA, Danila DC, Lin O, Gonzalez-Espinoza R, Gu B, Anand A, Smith K, Maslak P, Doyle GV, Terstappen LW, Lilja H, Heller G, Fleisher M, Scher HI. Circulating tumor cell analysis in patients with progressive castration-resistant prostate cancer. Clin Cancer Res. 2007 Apr 1;13(7):2023-9. doi: 10.1158/1078-0432.CCR-06-2701. PMID 17404082
- [Background] Zapatero A, Rios P, Marin A, Minguez R, Garcia-Vicente F. Dose escalation with three-dimensional conformal radiotherapy for prostate cancer. Is more dose really better in high-risk patients treated with androgen deprivation? Clin Oncol (R Coll Radiol). 2006 Oct;18(8):600-7. doi: 10.1016/j.clon.2006.06.010. PMID 17051950
- [Background] Moreno JG, Miller MC, Gross S, Allard WJ, Gomella LG, Terstappen LW. Circulating tumor cells predict survival in patients with metastatic prostate cancer. Urology. 2005 Apr;65(4):713-8. doi: 10.1016/j.urology.2004.11.006. PMID 15833514
- [Background] Fehm T, Sagalowsky A, Clifford E, Beitsch P, Saboorian H, Euhus D, Meng S, Morrison L, Tucker T, Lane N, Ghadimi BM, Heselmeyer-Haddad K, Ried T, Rao C, Uhr J. Cytogenetic evidence that circulating epithelial cells in patients with carcinoma are malignant. Clin Cancer Res. 2002 Jul;8(7):2073-84. PMID 12114406
- [Background] Zapatero A, Minguez R, Nieto S, Martin de Vidales C, Garcia-Vicente F. Post-treatment prostate biopsies in the era of three-dimensional conformal radiotherapy: what can they teach us? Eur Urol. 2009 Apr;55(4):902-9. doi: 10.1016/j.eururo.2008.04.076. Epub 2008 May 7. PMID 18485578
- [Background] Zapatero A, Garcia-Vicente F, Martin de Vidales C, Cruz Conde A, Ibanez Y, Fernandez I, Rabadan M. Long-term results after high-dose radiotherapy and adjuvant hormones in prostate cancer: how curable is high-risk disease? Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1279-85. doi: 10.1016/j.ijrobp.2010.07.1975. Epub 2010 Oct 6. PMID 20932659
- [Background] Olivier Gomez C, Carballido Rodriguez J. [Circulating tumor cells: isolation, quantification, and relevance of their translation into clinical practice]. Actas Urol Esp. 2010 Jan;34(1):3-5. No abstract available. Spanish. PMID 20223125
- [Background] Alix-Panabieres C, Riethdorf S, Pantel K. Circulating tumor cells and bone marrow micrometastasis. Clin Cancer Res. 2008 Aug 15;14(16):5013-21. doi: 10.1158/1078-0432.CCR-07-5125. PMID 18698019
- [Background] Mocellin S, Keilholz U, Rossi CR, Nitti D. Circulating tumor cells: the 'leukemic phase' of solid cancers. Trends Mol Med. 2006 Mar;12(3):130-9. doi: 10.1016/j.molmed.2006.01.006. Epub 2006 Feb 20. PMID 16488189
- [Background] Cabanes A, Vidal E, Aragones N, Perez-Gomez B, Pollan M, Lope V, Lopez-Abente G. Cancer mortality trends in Spain: 1980-2007. Ann Oncol. 2010 May;21 Suppl 3:iii14-20. doi: 10.1093/annonc/mdq089. PMID 20427355
- [Background] Ghossein RA, Bhattacharya S. Molecular detection and characterisation of circulating tumour cells and micrometastases in solid tumours. Eur J Cancer. 2000 Aug;36(13 Spec No):1681-94. doi: 10.1016/s0959-8049(00)00152-0. PMID 10959054
- [Background] Llanes L, Ferruelo A, Lujan M, Pascual C, Garcia-Mediero JM, Berenguer A. Quantitative real-time reverse transcription: polymerase chain reaction of prostate-specific antigen (PSA) for detection of circulating prostatic cells in patients with clinically localized prostate cancer. Prostate Cancer Prostatic Dis. 2005;8(3):248-52. doi: 10.1038/sj.pcan.4500801. PMID 15897916
- [Background] Zapatero A, Valcarcel F, Calvo FA, Algas R, Bejar A, Maldonado J, Villa S. Risk-adapted androgen deprivation and escalated three-dimensional conformal radiotherapy for prostate cancer: Does radiation dose influence outcome of patients treated with adjuvant androgen deprivation? A GICOR study. J Clin Oncol. 2005 Sep 20;23(27):6561-8. doi: 10.1200/JCO.2005.09.662. PMID 16170164
- [Background] Roach M 3rd, Hanks G, Thames H Jr, Schellhammer P, Shipley WU, Sokol GH, Sandler H. Defining biochemical failure following radiotherapy with or without hormonal therapy in men with clinically localized prostate cancer: recommendations of the RTOG-ASTRO Phoenix Consensus Conference. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):965-74. doi: 10.1016/j.ijrobp.2006.04.029. PMID 16798415
- [Background] Cristofanilli M. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. Semin Oncol. 2006 Jun;33(3 Suppl 9):S9-14. doi: 10.1053/j.seminoncol.2006.03.016. PMID 16797376
- [Background] Bolla M, Collette L, Van Tienhoven G, et al. Ten-year results of long-term adjuvant androgen deprivation with goserelin in patients with locally advanced prostate cancer treated with radiotherapy: A phase III EORTC study. Int J Radiat Oncol Biol Phys 2008;72:S30-S31.
- [Background] Resel Folkersma L, Olivier Gomez C, San Jose Manso L, Veganzones de Castro S, Galante Romo I, Vidaurreta Lazaro M, de la Orden GV, Arroyo Fernandez M, Diaz Rubio E, Silmi Moyano A, Maestro de Las Casas MA. Immunomagnetic quantification of circulating tumoral cells in patients with prostate cancer: clinical and pathological correlation. Arch Esp Urol. 2010 Jan-Feb;63(1):23-31. PMID 20157216
- [Result] Zapatero A, Gomez-Caamano A, Cabeza Rodriguez MA, Muinelo-Romay L, Martin de Vidales C, Abalo A, Calvo Crespo P, Leon Mateos L, Olivier C, Vega Piris LV. Detection and dynamics of circulating tumor cells in patients with high-risk prostate cancer treated with radiotherapy and hormones: a prospective phase II study. Radiat Oncol. 2020 Jun 1;15(1):137. doi: 10.1186/s13014-020-01577-5. PMID 32487218
- [Result] A. Zapatero, A. Gomez Caamaño, M. D. L. A. Cabeza Rodriguez, L. Muinelo-Romay, C. Martin de Vidales C, A. Abalo, et al. Monitoring of Circulating Tumor Cells in Patients With High-Risk Nonmetastatic Prostate Cancer Treated With Radiation Therapy and Hormones: Preliminary Data of an Observational Prospective Phase 2 Study. International Journal of Radiation Oncology • Biology • Physics, Vol. 99, Issue 2, E280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 patients included: 2 patients were not included in the final enrollment due to inegibility criteria
Groups:
- Circulating Prostatic Tumor Cells in the Peripheral Blood: Patients that satisfy inclusion criteria, and after signing informed consent, will extract 1 blood sample (7.5 mL):
  1. prior to any treatment;
  2. following AD and prior to RT; and
  3. following the end of RT (1-3 months afterwards).
  The quantification of CTC in blood samples will be done with the CellSearch® system.
Period: Overall Study
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Started | 66
Completed | 65
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- CTCs Analysis: Prospective analysis of biologic samples from PB of 65 patients with localized high-risk PCa (NCCN 2011) treated with RTC-3D-IMRT combined with ADT. Following the sign of the informed consent of the patient, the blood samples will be analyzed for CTCs using an immunomagnetic method based on the CellSearch system in 4 periods of time:
  1. Prior to any treatment (baseline- Time 1)
  2. Following ADT and prior to RT (Time 2)
  3. Following the end of RT (1-3 months afterwards) (Time 3)
  4. Following 9 -12 after RT in those cases in cases of one turn (+) in CTCs in the 2nd or 3rd determination
Arm/Group | CTCs Analysis
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 50
Age, Continuous [Median (Full Range); unit: years] | 71 [53 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 65
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 66
Median PSA (ng/mL) [Median (Full Range); unit: ng/mL] | 12.6 [3.2 to 68.7]
PSA pre-treatment [Count of Participants; unit: Participants]
  < 10 ng/mL | 24
  10 - 20 ng/mL | 19
  > 20 ng/mL | 23
Gleason score [Count of Participants; unit: Participants]
  Gleason sum =< 6 Better prognosis | 5
  Gleason sum = 7 | 33
  Gleason sum = 8 - 10 Worst prognosis | 28
Clinical T Stage according to AJCC seventh edition [Count of Participants; unit: Participants]
  T1 Best prognosis | 1
  T2 | 17
  T3 Worst prognosis | 48
Clinical N Stage according to AJCC seventh edition [Count of Participants; unit: Participants]
  N0 Best prognosis | 53
  N1 Worst prognosis | 13
Radiotherapy dose (Gy) [Median (Full Range); unit: Gy]
  3D Conformal RT | 76.3 [74.8 to 79.2]
  IMRT-IGRT | 81.7 [70.6 to 82.8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Circulating Tumor Cells in the Peripheral Blood
Description: Initially a cutoff point of > 1 or more circulating cells per 7.5 mL of blood will be taken as the reference baseline.
Time Frame: Basal
Measure: Count of Participants; unit: Participants
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Number analyzed (Participants) | 65
Participants
  Number of Participants with 0 CTCs | 60
  Number of Participants with =>1 CTCs | 5

2. Primary Outcome: Number of Participants With Circulating Tumor Cells in the Peripheral Blood
Description: (Initially a cutoff point of > 1 or more circulating cells per 7.5 mL of blood will be taken as the reference baseline).
Time Frame: Post-neoadjuvant hormone therapy and prior to radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Number analyzed (Participants) | 65
Participants
  Number of Participants with 0 CTCs | 54
  Number of Participants with =>1 CTCs | 8
  No Data | 3

3. Primary Outcome: Number of Participants With Circulating Tumor Cells in the Peripheral Blood
Description: (Initially a cutoff point of > 1 or more circulating cells per 7.5 mL of blood will be taken as the reference baseline).
Time Frame: Post-radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Number analyzed (Participants) | 65
Participants
  Number of Participants with 0 CTCs | 48
  Number of Participants with =>1 CTCs | 11
  No Data | 6

4. Primary Outcome: Number of Participants With Circulating Tumor Cells in the Peripheral Blood
Description: (Initially a cutoff point of > 1 or more circulating cells per 7.5 mL of blood will be taken as the reference baseline).
Time Frame: 9 - 12 months post-radiotherapy in cases with positivation after basal visit
Population: Patients with positivation after basal visit
Measure: Count of Participants; unit: Participants
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Number analyzed (Participants) | 13
Participants
  Number of Participants with 0 CTCs | 12
  Number of Participants with =>1 CTCs | 1

5. Secondary Outcome: Biochemical Failure-free Survival;
Description: Phoenix criteria (PSA Nadir +2 ng/mL)
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Number analyzed (Participants) | 65
Participants
  Yes | 64
  No | 1

6. Secondary Outcome: Overall Survival
Description: Defined as death due to any cause
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Number analyzed (Participants) | 65
Participants
  Yes | 59
  No | 6

7. Secondary Outcome: Metastasis-free Survival
Description: Defined as freedom from distant metastasis
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Number analyzed (Participants) | 65
Participants
  Yes | 64
  No | 1

8. Secondary Outcome: Cause Specific Survival
Description: Defined as death caused by prostate cancer
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
Number analyzed (Participants) | 65
Participants
  Yes | 65
  No | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Circulating Prostatic Tumor Cells in the Peripheral Blood
All-Cause Mortality (participants affected / at risk) | 7/65
Serious Adverse Events (participants affected / at risk) | 7/65
Other Adverse Events (participants affected / at risk) | 15/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circulating Prostatic Tumor Cells in the Peripheral Blood (N=65)
Postoperative of colon volvulus (Injury, poisoning and procedural complications) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Pneumomia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchoaspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastric GIST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ureter cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urethral estenosis (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circulating Prostatic Tumor Cells in the Peripheral Blood (N=65)
Late urinary symptoms Grade >= 2 (Renal and urinary disorders) | 9 (9)
Late rectal symptoms Grade >= 2 (Gastrointestinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT01800058/Prot_SAP_000.pdf